CLINICAL TRIAL: NCT06296563
Title: A Single Arm, Exploratory Clinical Study on the Perioperative Treatment of Resectable Intrahepatic Cholangiocarcinoma With the Combination of Adebrelimab and Apatinib and HAIC
Brief Title: Perioperative Treatment of Resectable Intrahepatic Cholangiocarcinoma With the Combination of Adebrelimab and Apatinib and HAIC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Lei ZHAO (Other)
Responsible Party: Sponsor-Investigator, Lei ZHAO, Director, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR1316-ICC-SD-001
Record Dates: First submitted 2024-02-28; First posted 2024-03-06 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Intrahepatic Cholangiocarcinoma
MeSH Terms: conditions — Cholangiocarcinoma | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HAIC+Adebrelimab+apatinib (Experimental): Neoadjuvant therapy with Adebrelimab combined with apatinib and FOLFOX-HAIC for 2 cycles (1 treatment cycle every 21 days, apatinib only used for the first cycle), and surgery was performed 14-28 days after the end of treatment. After 28 days of surgery, patients will continue to receive adjuvant treatment with Adebrelimab combined with apatinib.
  Interventions: Procedure: HAIC; Drug: Adebrelimab; Drug: Apatinib

INTERVENTIONS:
Procedure: HAIC — FOLFOX-hepatic artery infusion for 2 times.
Drug: Adebrelimab — Adebrelimab 1200mg, ivgtt, d1, q3w,up to one year of use at most.
Drug: Apatinib — Apatinib 250mg, po, qd,q3w,up to one year of use at most.

SUMMARY:
The goal of this clinical trial is to explore the efficacy and safety of combined infusion chemotherapy with Adebrelimab and Apatinib in the perioperative treatment of resectable intrahepatic cholangiocarcinoma patients. The main question it aims to answer are:

How to improve the survival of patients with intrahepatic cholangiocarcinoma and prolong the recurrence time after surgery.

Participants will receive receive neoadjuvant therapy with Adebrelimab combined with apatinib and FOLFOX-HAIC for 2 cycles (1 treatment cycle every 21 days, apatinib only used for the first cycle), and surgery was performed 14-28 days after the end of treatment. After 28 days of surgery, patients will continue to receive adjuvant treatment with Adebrelimab combined with apatinib for a maximum of one year.

ELIGIBILITY:
Inclusion Criteria:

* 1. Pathological diagnosis as malignant tumor of Intrahepatic Cholangiocarcinoma;
* 2. According to the UICC/AJCC TNM staging system (8th edition, 2017), resectable subjects were classified as Ib-IIIb stages;
* 3. aged ≥ 18 years at the time of signing the Informed consent form (ICF);
* 4. Expected survival time>3 months;
* 5. Both men and women are eligible;
* 6. The patient's Eastern Oncology Collaborative Group (ECOG) physical condition score is 0 or 1;
* 7. No serious complications, such as hypertension, coronary heart disease, or history of mental illness, and no history of severe allergies; Non pregnancy and non lactation period;
* 8. The organ and blood system functions of the subjects meet the following requirements:

  1. Absolute neutrophil count (ANC) ≥ 1.5 × 10 ^ 9/L;
  2. Platelet count ≥ 75 × 10 ^ 9/L;
  3. Hemoglobin ≥ 90 g/L;
  4. Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN);
  5. Aspartate aminotransferase (AST) and alanine aminotransferase ≤ 2.5 x ULN;
  6. Albumin ≥ 3g/dL
  7. Creatinine ≤ 1.5 x ULN
* 9. The subjects can understand and sign the informed consent form to participate in the experimental study; Good compliance.
* 10. Participants who have not undergone any local or systemic treatment for tumors in the past, and have undergone radical resection surgery for biliary tract cancer before recurrence for at least 2 years, can be included;
* 11. Subjects with potential fertility need to use a medically approved contraceptive measure (such as an intrauterine device, contraceptive pill, or condom) during the study treatment period and within one month after the end of the study treatment period; And within 72 hours before enrollment, the serum or urine HCG test must be negative and must be non lactating;

Exclusion Criteria:

* 1. Patients who received PD-1, PD-L1, PD-L2, or CTLA-4 inhibitors before enrollment, or patients who directly received another stimulating or co inhibitory T cell receptor (such as CTLA-4, CD137);
* 2. Use any other investigational drugs within 4 weeks prior to enrollment;
* 3. Any history of active autoimmune diseases or autoimmune diseases (such as interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, myocarditis, nephritis, hyperthyroidism, hypothyroidism after hormone replacement therapy); Children with asthma who have completely improved in adulthood and do not require any intervention can be included, but patients who require intervention with bronchodilators cannot be included;
* 4. Congenital or acquired immunodeficiency, such as infection with human immunodeficiency virus (HIV), active hepatitis B (HBV DNA 500IU/ml), hepatitis C (hepatitis C antibody positive, HCV-RNA above the detection limit of the analysis method), or co infection with hepatitis B and hepatitis C;
* 5. Serious infection (such as intravenous infusion of antibiotics, antifungal or antiviral drugs) occurred within 4 weeks before the first administration, or unexplained fever>38.5 ° C occurred during screening/before the first administration;
* 6. History of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* 7. Suffering from uncontrollable mental illness;
* 8. The simultaneous occurrence of serious and/or uncontrollable diseases may affect the participation of the study, such as unstable angina pectoris, myocardial infarction within 6 months, unstable symptomatic arrhythmia, symptomatic congestive heart failure, poorly controlled diabetes, serious activities, uncontrollable infection after insufficient biliary drainage (such as tumor blocking the bile duct);
* 9. Pregnancy (positive pregnancy test) or lactation period;
* 10. Other cancers that have occurred in the past (within the past 5 years) or simultaneously, excluding non melanoma skin cancer and in situ cancer;
* 11. History of allergy or hypersensitivity to any investigational drug;
* 12. Currently abusing alcohol or illegal drugs;
* 13. Unable or unwilling to sign informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Pathologic complete response (pCR) | Up to one year
  The proportion of subjects whose postoperative pathological examination did not detect residual cancer cells.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to one year
  Objective response rate
Event free survival (EFS) | Up to two years
  The time from enrollment to the scheduled occurrence of events, including death, disease recurrence, disease progression, etc
Overall Survival (OS) | Up to two years
  Overall Survival：The survival time from enrollment to death from any cause.
Disease Control Rate (DCR) | Up to one year
  Disease Control Rate: Ratio of complete response (CR)+partial response (PR)+stable disease (SD)

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No